CLINICAL TRIAL: NCT01590264
Title: rTMS Bimodal Treatment For Patients With Subjective Idiopathic Tinnitus: A Pilot Study
Brief Title: rTMS Bimodal Treatment For Tinnitus: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor, Director of Clinical Outcomes, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201204069
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2012-09

CONDITIONS: Tinnitus
Keywords: tinnitus; bimodal stimulation; rTMS; Repetitive Transcranial Magnetic Stimulation
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bimodal rTMS (Other): Open-label and single-arm rTMS bimodal treatment with placement of magnet over Dorsolateral Prefrontal Cortex (DLPFC) and Temporoparietal Junction (TPJ) for 2 weeks of treatment (10 days)
  Stimulation Settings:
  DLPFC Stimulation Frequency 10 Hz Intensity 110% of motor threshold On 5 seconds Off 15 seconds Total Trains 80 per session Total pulses session 4000/session Duration session 26.6 minutes Total pulses (study) 40000
  TPJ Stimulation Frequency 1 Hz Intensity 110% of motor threshold On 900 seconds Off 60 seconds Total Trains 2 per session Total Pulses session 1800 Duration session 31 minutes Total Pulses study 18000
  Interventions: Device: Bimodal rTMS

INTERVENTIONS:
Device: Bimodal rTMS — High frequency (10 Hz) at 110% of the motor threshold TMS delivered over the left dorsolateral prefrontal cortex, subsequently, a low frequency TMS (1 Hz) at 110% motor threshold will be delivered over 31 minutes over the TPJ area, according to the protocol below.
  DLPFC Stimulation Frequency 10 Hz Intensity 110% of motor threshold On 5 seconds Off 15 seconds Total Trains 80 per session Total pulses session 4000/session Duration session 26.6 minutes Total pulses (study) 40000
  TPJ Stimulation Frequency 1 Hz Intensity 110% of motor threshold On 900 seconds Off 60 seconds Total Trains 2 per session Total Pulses session 1800 Duration session 31 minutes Total Pulses study 18000
  Other Names: The rTMS system is a Magpro R 30 stimulator.

SUMMARY:
Repetitive Transcranial Magnetic Stimulation (rTMS) is a novel brain stimulation technique that uses pulsating magnetic fields to stimulate underlying neurons in the cerebral cortex. The investigators propose an open-label pilot study investigating the effectiveness of rTMS in the treatment of tinnitus stimulation of the left dorsolateral prefrontal cortex (DLPFC), an area known to be important for mood and attention, along with stimulation of the left temporoparietal cortex (TPC). This is a feasibility pilot study.

DETAILED DESCRIPTION:
Converging data implicate structures of the brain that are important for mood and attention as playing a role in the maintenance of tinnitus; suggesting an alternative rTMS treatment approach that targets these structures. A growing number of studies demonstrate involvement of the prefrontal cortex in the generation and maintenance of tinnitus. rTMS stimulation in the dorsolateral prefrontal cortex in association with stimulation in the temporoparietal cortex has been shown to increase the durability of the TPC stimulation. The independent effect of rTMS stimulation to the DLPFC is not known. Studies in depression suggest that increasing the intensity and duration of stimulation has beneficial treatment effects. However, the field is new and more work is needed to assess the effectiveness of this treatment, predictors and correlates of response, and safety.

Recent exciting work in schizophrenia used a bimodal (DLPFC and TPC) treatment approach in pharmacologically non-responsive patients. The study used high-frequency stimulation to the left DLPFC and low-frequency stimulation to the left TPC. Bimodal rTMS stimulation of left DLPFC and left TPC induced clinical improvement in pharmacologically non-responsive schizophrenia patients and may have improved their short-term verbal memories.57

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 60 years.
* Subjective, idiopathic, troublesome, unilateral or bilateral, non-pulsatile tinnitus of ≥ 2 month's duration but no greater than 5 year's duration.
* Bothersome Tinnitus according to Tinnitus Handicap Inventory score.
* Must be able to understand, speak, read and write English proficiently
* Able to provide informed consent
* Women who are of childbearing potential must agree to use a medically acceptable form of birth control and must have a negative urine pregnancy test at screening

Exclusion Criteria:

* •• Patients with tinnitus related to cochlear implantation, retrocochlear lesion, or other known anatomic/structural lesions of the ear and temporal bone. Patients with a history of stapedectomy and insertion of implant will be excluded.

  * Hypersensitive to noises (hyperacusis)
  * Patients with history of head injury with 15 minutes or more loss of consciousness or required medical treatment.
  * Patients with cardiac pacemakers; intracardiac lines; implanted medication pumps; implanted electrodes in the brain; other implanted electrical or magnetic medical devices; or other intracranial metal objects or shrapnel, with the exception of dental fillings.
  * Patients with additional significant neurological disorders including increased intracranial pressure, brain mass, epileptic seizures (or family history of epileptic seizures), history of stroke, transient ischemic attack within 2 years, cerebral aneurysm, Huntington's chorea or multiple sclerosis.
  * Patients with an acute or unstable medical condition including all patients with any significant heart disease, pneumonia, uncontrolled hypertension, or other disorders which would require stabilization prior to initiation of transcranial magnetic stimulation.
  * Active alcohol and/or drug dependence or history of alcohol and/or drug dependence within the last year.
  * Patients with moderate to severe clinical depression as evidenced by a score of 15 or greater on the PHQ-9.
  * Patients who, in the opinion of the psychiatric sub-investigator, demonstrate moderate to severe depressive symptoms according to DSM-IV-TR criteria for Major Depressive Disorder.
  * Patients with psychiatric illness or trauma which would prohibit participation in the study.
  * Patients with active psychotic symptoms or a history of psychotic disorder
  * Female patients of child-bearing potential, unless sterilized or using an appropriate form of birth control acceptable to the research team.
  * Currently breastfeeding
  * Currently pregnant
  * Patients will be excluded if a motor threshold cannot be elicited,
  * Patients whose ability to give informed consent is in question
  * Undiagnosed symptomatic hypertension: .
  * Undiagnosed asymptomatic hypertension:
  * Any patient who has scheduled an elective surgery or change in medication during the 5 weeks of the study.
  * Use of Neuromonics Device during duration of study or currently in Tinnitus Retraining Program during course of study.
  * Any medical condition that, in the opinion of the investigators, confounds study results or places the subject at greater risk.
  * Patients currently taking psychotropic medications including antidepressants, benzodiazepines, anticonvulsants, stimulants, antipsychotics, or anxiolytics.
  * Tinnitus related to a Workman's Compensation claim or litigation-related event that is still pending.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine, St. Louis
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Burton H, Wineland A, Bhattacharya M, Nicklaus J, Garcia KS, Piccirillo JF. Altered networks in bothersome tinnitus: a functional connectivity study. BMC Neurosci. 2012 Jan 4;13:3. doi: 10.1186/1471-2202-13-3. PMID 22217183
- [Background] Piccirillo JF, Garcia KS, Nicklaus J, Pierce K, Burton H, Vlassenko AG, Mintun M, Duddy D, Kallogjeri D, Spitznagel EL Jr. Low-frequency repetitive transcranial magnetic stimulation to the temporoparietal junction for tinnitus. Arch Otolaryngol Head Neck Surg. 2011 Mar;137(3):221-8. doi: 10.1001/archoto.2011.3. PMID 21422304
- [Background] Pierce KJ, Kallogjeri D, Piccirillo JF, Garcia KS, Nicklaus JE, Burton H. Effects of severe bothersome tinnitus on cognitive function measured with standardized tests. J Clin Exp Neuropsychol. 2012;34(2):126-34. doi: 10.1080/13803395.2011.623120. Epub 2011 Dec 14. PMID 22168528
- [Background] Oh SY, Kim YK. Adjunctive treatment of bimodal repetitive transcranial magnetic stimulation (rTMS) in pharmacologically non-responsive patients with schizophrenia: a preliminary study. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Dec 1;35(8):1938-43. doi: 10.1016/j.pnpbp.2011.07.015. Epub 2011 Aug 5. PMID 21840364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from Washington University Otolaryngology and Audiology clinics.
Pre-assignment Details: Subjects were enrolled for one pre-treatments screening visits, received two weeks of rTMS treatment, and were assessed at the last treatment day. There was no additional follow-up.
Period: Overall Study
Arm/Group | Bimodal rTMS
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bimodal rTMS
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Subject will be queried for Adverse Events daily for 2 weeks of treatment. This is foremost a feasibility study, so measure of Adverse Events and relation to treatment is primary outcome.
Time Frame: Daily for 2 weeks.
Population: Pilot study based on convenience sample.
Measure: Number; unit: participants
Arm/Group | Bimodal rTMS
Number analyzed (Participants) | 5
participants | 0

2. Secondary Outcome: Change in Tinnitus Handicap Inventory
Description: Participant will complete the Tinnitus Handicap Inventory (THI)at the end of 2 weeks of treatment. Difference of the THI post treatmement minus baseline THI was calculated. Scale ranges in scores from 0 to 100 with 0 = no bother and 100 being the most bothered.
Time Frame: Baseline, 2 weeks
Population: Pilot study convenience sample
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Bimodal rTMS
Number analyzed (Participants) | 5
units on a scale | -12 [-26 to 0]

ADVERSE EVENTS:
Arm/Group | Bimodal rTMS
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes